CLINICAL TRIAL: NCT01253681
Title: A Phase 1b Open-Label, Multi-Center Study of AMG 386 in Combination With Paclitaxel and Carboplatin in Subjects With High-Risk Stage I and Stages II-IV Epithelial Ovarian, Primary Peritoneal or Fallopian Tube Cancers
Brief Title: Study of AMG 386 in Combination With Paclitaxel and Carboplatin in Subjects With Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20090155
Record Dates: First submitted 2010-10-21; First posted 2010-12-03 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Carcinoma; Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cancer
Keywords: AMG 386; Ovarian Cancer
MeSH Terms: conditions — Carcinoma; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — trebananib; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AMG 386, paclitaxel and carboplatin (Experimental): 15 mg/Kg AMG 386 IV (intravenous) weekly plus paclitaxel and carboplatin IV Q3W for 18 weeks, followed by 15mg/Kg AMG 386 IV (intravenous) weekly alone for an additional 18 months.
  Interventions: Drug: AMG 386, paclitaxel and carboplatin

INTERVENTIONS:
Drug: AMG 386, paclitaxel and carboplatin — 15 mg/Kg AMG 386 IV (intravenous) weekly plus paclitaxel and carboplatin IV Q3W for 18 weeks, followed by 15mg/Kg AMG 386 IV (intravenous) weekly alone for an additional 18 months.

SUMMARY:
To evaluate whether AMG 386 in combination with paclitaxel and carboplatin is safe and well tolerated in the first-line treatment of high-risk stage I and stages II-IV epithelial ovarian, primary peritoneal and fallopian tube cancers. The hypothesis is that AMG 386 in combination with carboplatin and paclitaxel is safe and well tolerated.

DETAILED DESCRIPTION:
To evaluate whether AMG 386 in combination with paclitaxel and carboplatin is safe and well tolerated in the first-line treatment of high-risk stage I and stages II-IV epithelial ovarian, primary peritoneal and fallopian tube cancers. The hypothesis is that AMG 386 in combination with carboplatin and paclitaxel is safe and well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects more than 18 years of age with newly diagnosed high-risk FIGO Stage I (grade 3, or aneuploid grade 1 or 2) or Stages II-IV epithelial ovarian, primary peritoneal and fallopian tube cancer with an indication for first-line treatment with paclitaxel and carboplatin x 6 cycles. Subjects with pseudomyxoma, mesothelioma, adenocarcinoma of unknown primary tumor, sarcoma, or neuroendocrine histology are excluded.
* Subjects with high-risk stage I, stage II, or stage IIIA-B must have had prior primary debulking surgery that occurred no less than 4 weeks, and no more than 12 weeks, prior to enrollment. Subjects must have recovered fully from surgery in the opinion of the investigator
* Subjects with Stage IIIC or IV disease who have not had primary debulking surgery must have planned interval debulking surgery following 3 cycles of AMG 386, paclitaxel and carboplatin
* Female 18 years of age or older at the time the written informed consent is obtained
* Subjects of child-bearing potential who have not undergone a bilateral salpingo-oophorectomy and are sexually active must consent to use an accepted and effective non-hormonal method of contraception (i.e, double barrier method (eg, condom plus diaphragm) from signing the informed consent through 6 months after last dose of study drug
* GOG Performance Status of 0 or 1
* Life expectancy ≥ 3 months (per investigator opinion)
* Subject plans to begin protocol-directed therapy within 7 days from enrollment
* Adequate organ and hematological function as evidenced by the following laboratory studies prior to enrollment:

Hematological function, as follows:

* Hemoglobin ≥ 9 g/dL
* Absolute neutrophil count (ANC) ≥ 1.5 x 10x9/L
* Platelet count ≥ 100 x 10x9/L and ≤ 850 x 10x9/L
* PTT or aPTT ≤ 1.5 x ULN per institutional laboratory range and INR ≤ 1.5

Renal function, as follows:

* Urinary protein quantitative value of ≤ 30 mg/dL in urinalysis or ≤ 1+ on dipstick, unless quantitative protein is < 1000 mg in a 24 hour urine sample
* Creatinine clearance > 40 mL/min per 24-hr urine collection or calculated according to the Cockcroft-Gault formula

Hepatic function, as follows:

* AST and ALT ≤ 2.5 x ULN per institutional laboratory range (or ≤ 5 x ULN if liver metastases are present)
* Total bilirubin ≤ 1.5x institutions' ULN Nutritional
* Albumin ≥ 2.8 g/dL

Exclusion Criteria:

* Prior use of anticancer therapy or experimental therapy for epithelial ovarian, primary peritoneal or fallopian tube cancers
* Previous abdominal and/or pelvic external beam radiotherapy
* Subjects believed to be a higher than average risk of bowel perforation. This includes current symptoms of partial or complete bowel obstruction, recent (within 6 months) history of fistula or bowel perforation, subjects requiring total parenteral nutrition and continuous hydration
* History of arterial or venous thromboembolism within 12 months prior to enrollment
* History of clinically significant bleeding within 6 months prior to enrollment
* History of central nervous system metastasis
* Known active or ongoing infection (except uncomplicated urinary tract infection) within 14 days prior to enrollment
* Currently or previously treated with AMG 386, or other molecules that inhibit the angiopoietins or Tie2 receptor
* Current or within 30 days prior to enrollment treatment with immune modulators such as systemic cyclosporine or tacrolimus
* Prior myeloablative high-dose chemotherapy with allogeneic or autologous stem cell (or bone marrow) transplant
* Clinically significant cardiac disease within 12 months prior to enrollment, including myocardial infarction, unstable angina, grade 2 or greater peripheral vascular disease, cerebrovascular accident, transient ischemic attack, congestive heart failure, or arrhythmias not controlled by outpatient medication or placement of percutaneous transluminal coronary angioplasty/stent
* Uncontrolled hypertension as defined as diastolic blood pressure > 90 mmHg OR systolic blood pressure > 140 mmHg. The use of anti-hypertensive medications to control hypertension is permitted
* Subjects with a history of prior malignancy, except:

Malignancy treated with curative intent and with no known active disease present for ≥ 3 years prior to enrollment and felt to be at low risk for recurrence by treating physician, Adequately treated non-melanomatous skin cancer or lentigo maligna without evidence of disease Adequately treated cervical carcinoma in situ without evidence of disease

* Major surgery within 28 days prior to enrollment or still recovering from prior surgery
* Minor surgical procedures, including placement of tunneled central venous access device, within 3 days prior to enrollment
* History of allergic reactions to bacterially-produced proteins
* Hypersensitivity to paclitaxel or drugs using the vehicle cremophor
* Pregnant (ie, positive beta-human chorionic gonadotropin test) or is breast feeding or planning to become pregnant within 6 months after the end of treatment
* Subject has known positive test(s) for human immunodeficiency virus (HIV) infection, hepatitis C virus, acute or chronic active hepatitis B infection
* Any condition which in the investigator's opinion makes the subject unsuitable for study participation
* Any uncontrolled concurrent illness or history of any medical condition that may interfere with the interpretation of the study results
* Non-healing wound, ulcer (including gastrointestinal) or fracture
* Subject has previously been enrolled onto this study
* Subject will not be available for follow-up assessment
* Subject has known sensitivity to any of the products to be administered during dosing
* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-11; Primary Completion 2012-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
To evaluate whether AMG 386 in combination with paclitaxel and carboplatin is safe and well tolerated in the first-line treatment of high-risk stage I and stages II-IV epithelial ovarian, primary peritoneal and fallopian tube cancers. | 18 weeks of combination therapy

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics (Cmax, AUC and Cmin) of AMG 386 in combination with carboplatin and paclitaxel | Week 1 until Week 7
To estimate the incidence of anti-AMG 386 antibody formation | Week 1 until maximum of 1 year following first dose
To evaluate the objective response rate (ORR) among subjects receiving AMG 386 in combination with carboplatin and paclitaxel | From date of first dose until the subject reaches End of Study. This will continue until 36 months after the last subject has been enrolled.
To evaluate the duration of response (DOR) among subjects receiving AMG 386 in combination with carboplatin and paclitaxel | From date of first dose until the subject reaches End of Study. This will continue until 36 months after the last subject has been enrolled.
To evaluate progression-free survival (PFS) among subjects receiving AMG 386 in combination with carboplatin and paclitaxel | From date of first dose until the subject reaches End of Study. This will continue until 36 months after the last subject has been enrolled.
To evaluate the number of participants with adverse events and clinical laboratory abnormalities | 96 weeks
To evaluate the effect of AMG 386 on the pharmacokinetics (Cmax, AUC and Cmin) of carboplatin and paclitaxel | Week 1 until Week 7

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (7):
- Australia (3):
  - Research Site, Footscray, Victoria
  - Research Site, Malvern, Victoria
  - Research Site, Parkville, Victoria
- Belgium (2):
  - Research Site, Brussels
  - Research Site, Leuven
- Spain (2):
  - Research Site, Barcelona, Catalonia
  - Research Site, Madrid, Madrid

REFERENCES:
- [Derived] Vergote I, Oaknin A, Baurain JF, Ananda S, Wong S, Su X, Wu B, Zhong Z, Warner D, Casado A. A phase 1b, open-label study of trebananib in combination with paclitaxel and carboplatin in patients with ovarian cancer receiving interval or primary debulking surgery. Eur J Cancer. 2014 Sep;50(14):2408-16. doi: 10.1016/j.ejca.2014.06.010. Epub 2014 Jul 15. PMID 25037684
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com